CLINICAL TRIAL: NCT03848507
Title: Impact of Hyperoncotic Albumin to Support Blood Loss Replacement on Plasma Volume Expansion in Cystectomy Patients.
Brief Title: Impact of Hyperoncotic Albumin to Support Blood Loss Replacement
Acronym: HYPALB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPALB
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Blood Loss, Surgical; Fluid Retention
Keywords: hyperoncotic albumin, blood loss, fluid replacement, cystectomy
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20% Albumin (Experimental): Administration of 3ml per kg bodyweight of 20% albumin within 30 min during cystectomy.
  Interventions: Drug: albumin 20%

INTERVENTIONS:
Drug: albumin 20% — Intravenous administration of 20% albumin during cystectomy

SUMMARY:
Fluid treatment is usually performed with either balanced crystalloid fluids or iso-oncotic colloids, (synthetic colloids, plasma and 5% albumin). Doubts have been raised about synthetic colloids (impairment of renal function and coagulation), and the natural albumin has been used more extensively. Albumin is the main protein responsible for plasma oncotic pressure and its volume expansion effect. An alternative therapeutic option is the mobilization of tissue fluid by infusing a small amount of hyper-oncotic fluid like the 20% albumin solution (endogenous fluid recruitment).

The primary objective of this study is to test the effect of 20% albumin on plasma volume expansion and fluid recruitment in the frame of blood loss replacement during cystectomy using established fluid kinetic models.

The investigators expect that fluid replacement with crystalloid will be better sustained intravascularly with the administration of 20% albumin and be able to recruit fluid into the vascular compartment.

DETAILED DESCRIPTION:
Bladder cancer occurs mainly in old comorbid patients. The standard treatment of localized muscle invasive bladder cancer is pelvic lymph node dissection and open radical cystectomy with urinary diversion. Optimal perioperative fluid management for this surgery is challenging and still controversial in terms of how much to perfuse, choice of fluids (crystalloids and colloids) to restore hydrated state and volemia.

Fluid treatment is usually performed with either balanced crystalloids fluids or iso-oncotic synthetic colloids, plasma or 5% albumin. Because crystalloids quickly equilibrate between the intravascular and interstitial volumes, they are mainly used to treat dehydration and temporary volume deficits. Iso-oncotic colloids remain intravascular for a prolonged period. Doubts have been raised about synthetic colloids, and the natural albumin has been used more extensively. Albumin is the main protein responsible for plasma oncotic pressure and its volume expansion effect. An alternative therapeutic option is the mobilization of tissue fluid by infusing a small amount of hyper-oncotic fluid like the 20% albumin solution (endogenous fluid recruitment).

There are still unknown aspects of the physiological effects of hyper-oncotic albumin. One of them is the, in this study investigated, effect of 20% albumin on plasma volume expansion, fluid recruitment, and crystalloid kinetic in the frame of blood loss replacement during cystectomy.

It is expected that fluid replacement with crystalloid will be better sustained intravascularly with the administration of 20% albumin.

ELIGIBILITY:
Inclusion Criteria:

* Non emergent radical cystectomy with urinary diversion
* Adult: older than 18 years
* Written informed consent

Exclusion Criteria:

* Significant renal dysfunction: glomerular filtration rate < 60 ml/min/1,73 m² (Kidney Disease Outcomes Quality Initiative stage 3 or more )
* History of heart failure
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Women who are pregnant or breast feeding (exclusion of surgery per se)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Plasma volume expansion | 5 hours
  Calculated by kinetics models

SECONDARY OUTCOMES:
Colloid osmotic pressure | 5 hours
  Measured by oncometer
Fluid balance | 24 hours
  Composite score calculated according to fluid administered (crystalloid, colloids, blood products) and fluid loss (urine and blood)
Complications rate | 90 days
  Assessment of all complications occurring from postoperative day 1 to 90 according to the Clavien Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wuethrich, MD, Principal Investigator — Inselspital Bern Switzerland
Locations (1):
- Patrick Wuethrich, Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hahn RG, Wuethrich PY, Zdolsek JH. Can perioperative hemodilution be monitored with non-invasive measurement of blood hemoglobin? BMC Anesthesiol. 2021 May 6;21(1):138. doi: 10.1186/s12871-021-01351-4. PMID 33957864
- [Derived] Loffel LM, Hahn RG, Engel D, Wuethrich PY. Intraoperative Intravascular Effect of Lactated Ringer's Solution and Hyperoncotic Albumin During Hemorrhage in Cystectomy Patients. Anesth Analg. 2021 Aug 1;133(2):413-422. doi: 10.1213/ANE.0000000000005173. PMID 32947291